CLINICAL TRIAL: NCT01376427
Title: PROTOCOL TREATMENT for Acute Lymphoblastic Leukemia Ph '(BCR / ABL) POSITIVE PATIENTS AGED> 55 YEARS
Brief Title: Treatment of Acute Lymphoblastic Leukemia Ph '(BCR / ABL) Positive Patients Aged > 55 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-07OPH
Record Dates: First submitted 2011-06-02; First posted 2011-06-20 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphoblastic Leukemia Ph Positive
MeSH Terms: interventions — Dexamethasone; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone
Drug: Methotrexate — Methotrexate
Drug: Vincristine — Vincristine

SUMMARY:
This study proposes to provide adequate treatment and is based on current scientific evidence for elderly patients with ALL Bcr / Abl positive.

To determine whether low-dose chemotherapy associated with imatinib or dasatinib has acceptable tolerability in elderly patients.

To determine whether this association can increase the rate and quality of referrals to the results of the literature of imatinib as monotherapy for elderly patients

DETAILED DESCRIPTION:
Prephase (days -5 to -1) Dexamethasone 10 mg/m2 bolus day EV for 5 days (-5 to -1).

Intrathecal treatment (diagnosis and prophylactic / therapeutic) -5 days:

Methotrexate 12 mg

Systemic treatment:

* Imatinib 400 mg daily and continuous VO.
* Vincristine (VCR) 1 mg (absolute dose) EV 1, 8, 15 and 22.
* Dexamethasone (DEX): 10 mg/m2 EV, IM or PO days 1-2, 8-9 days 15-16, 22-23. .

Intrathecal chemotherapy:

Triple therapy was administered with methotrexate (MTX), cytosine arabinoside (ARA-C) and hydrocortisone, days 1, 8, 15 and 22 (five doses total prophylactic between prophase and induction):

MTX 12 mg ARA-C 40 mg Dexamethasone 4 mg

Maintenance during the first year will start after full recovery after induction and after complete reassessment of the disease (including mielograma and Bcr-Abl/Abl or Bcr-Abl/Gus ratio in peripheral blood) and will last until one year from the time of complete remission.

The basic treatment included imatinib 400 mg / day (or dasatinib), mercaptopurine at doses of 50 mg/m2 PO day and methotrexate 20 mg/m2 IM weekly.

One week every 3 months maintenance treatment added a "mini-reinduction" consisting

* VCR: 1 mg (absolute dose), i.v., day 1.
* Dexamethasone 40 mg / day, i.v. or p.o., days 1-2.
* not considered more doses of triple intrathecal therapy. Reinduction only be practiced during the first year after remission, so a total of 4 quarterly.

Maintenance treatment of second year

After the first year of maintenance will perform a complete reassessment of the disease (including myelogram) and if the patient remains in complete remission maintenance will continue (without reinduction) until two years from the time of diagnosis.

Maintenance treatment of third year During the third year after complete remission imatinib administered alone (or dasatinib

ELIGIBILITY:
Inclusion Criteria:

Adults over 55 years diagnosed with acute lymphoblastic leukemia Ph 'positive (Bcr / Abl positive) and previously untreated

Exclusion Criteria:

1. Other LAL negative for t (9; 22) and Bcr / Abl.
2. biphenotypic acute leukemias or bilinear with t (9; 22).
3. blast crisis of chronic myeloid leukemia progression during or after polychemotherapy treatment (including allo-BMT) or with inhibitors of tyrosine kinases.

   The criteria for exclusion from treatment (but not patient record) any of the following
4. General condition affected (grades 3 and 4 WHO scale), not attributable to the LAL.
5. Lack of consent by the patient to use their clinical d

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of response rate | 5 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events treated with chemotherapy and dasatinib combination | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol and all Hospital Pethema, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Ribera JM, Garcia O, Fernandez-Abellan P, Lavilla E, Bernal MT, Gonzalez-Campos J, Brunet S, Monteserin MC, Montesinos P, Sarra J, Calbacho M, Alvarez-Larran A, Tormo M, Oriol A; PETHEMA Group. Lack of negative impact of Philadelphia chromosome in older patients with acute lymphoblastic leukaemia in the thyrosine kinase inhibitor era: comparison of two prospective parallel protocols. Br J Haematol. 2012 Nov;159(4):485-8. doi: 10.1111/bjh.12043. Epub 2012 Sep 12. No abstract available. PMID 22966847
- See also: Related Info — https://www.fundacionpethema.es/